CLINICAL TRIAL: NCT05378100
Title: Low-Dose Ketamine Infusion for the Treatment of Multiple Sclerosis Fatigue (INKLING-MS)
Brief Title: Ketamine for Multiple Sclerosis Fatigue
Acronym: INKLING-MS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00322473
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis Fatigue
MeSH Terms: interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine-Ketamine (Experimental): Participants in this arm will receive two infusions of ketamine four weeks apart.
  Interventions: Drug: Ketamine
- Ketamine-Midazolam (Experimental): Participants in this arm will receive one infusion of ketamine followed four weeks later by an infusion of midazolam.
  Interventions: Drug: Ketamine; Drug: Midazolam
- Midazolam-Ketamine (Experimental): Participants in this arm will receive one infusion of midazolam followed four weeks later by an infusion of ketamine.
  Interventions: Drug: Ketamine; Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Infusion of ketamine 0.5 mg/kg over 40 minutes
Drug: Midazolam — Infusion of midazolam 0.05 mg/kg over 40 minutes
  Arms: Ketamine-Midazolam; Midazolam-Ketamine

SUMMARY:
The proposed study is a single-center, phase II, randomized, double-blind, parallel-group, active-placebo-controlled trial of intravenous low-dose ketamine in patients with MS fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a man or woman, 18 to 65 years of age, inclusive.
* Subject must be medically stable based on physical examination, medical history, and vital signs
* Subject must meet McDonald 2017 diagnostic criteria for multiple sclerosis based on the PI review of the medical records
* Subject must complain from fatigue as one of their main symptoms and have a screening MFIS score equal or higher than the cutoff based on gender, age, and education displayed in Table-226
* Subject must be ambulatory (able to walk at least 20 feet using bilateral assistance)
* Subject must have internet and email access and ability to use a computer or tablet or smartphone
* Subjects that are currently taking medication for alleviating fatigue (such as amantadine, modafinil and armodafinil, and amphetamine-like psychostimulants) at Screening are eligible to participate unless the medication is one of the disallowed therapies (Table 3). Subjects taking a fatigue medication at the Screening visit must have been receiving a stable dose for at least four weeks before the Screening visit and be willing to continue the medication at the same dose for the duration of the study.

Exclusion Criteria:

* BDI-II score of more than 29 (indicating severe depression)
* Having a known clear cause for secondary fatigue, such as untreated sleep apnea, untreated hypothyroidism, chronic liver disease, history of moderate to severe anemia (hemoglobin concentration of less than 9 gr/dl in men or less than 8 gr/dl in women).
* Neurodegenerative disorders other than relapsing or progressive MS
* Breastfeeding or pregnant
* History of coronary artery disease or congestive heart failure
* Uncontrolled hypertension at Screening (history of high blood pressure and screening systolic blood pressure >160 or diastolic blood pressure>100)
* History of severe liver disease, including cirrhosis
* Terminal medical conditions
* Currently treated for active malignancy
* Alcohol or substance abuse in the past year (except marijuana or other cannabinoids)
* A history of intolerance or allergic or anaphylactic reaction to ketamine or midazolam
* Clinically unstable medical or psychiatric disorders that require acute treatment as determined by the PI
* History of severe or untreated coronary artery disease or history of congestive heart failure
* History of prior ischemic or hemorrhagic stroke and cerebral vascular aneurysms.
* History of recurrent seizures or epilepsy
* Taking any disallowed therapy(ies), as noted in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) Score | Baseline (infusion visit) through four weeks after the infusion.
  The total score of the MFIS ranges from 0 to 84. Higher scores denote more severe fatigue.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | Baseline (infusion visit) through four weeks after the infusion.
  The total score of the FSS ranges from 1 to 7. Higher scores denote more severe fatigue.
Epworth Sleepiness Scale (ESS) | Baseline (infusion visit) through four weeks after the infusion.
  The total score of the ESS ranges from 0 to 24. Higher scores denote more severe sleepiness.
Beck Depression Inventory-II (BDI-II) | Baseline (infusion visit) through four weeks after the infusion.
  The total score of the BDI-IIranges from 0 to 63. Higher scores denote more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Bardia Nourbakhsh, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study and publication of key findings, the study investigators will make Final Research Data available to researchers upon written request. Researchers must adhere to a data sharing agreement. This agreement requires users to:
  (1) use the data only for research purposes; (2) not share the data with unauthorized users; (3) ensure that the data are protected from unauthorized persons; (4) require that the data be returned or destroyed at the end of the analysis; (5) provide certification of IRB review and approval.
Supporting Information: Study Protocol, SAP